CLINICAL TRIAL: NCT03823846
Title: The Effect of Doctor-nurse-patient Cooperative Analgesic Linkage Program on Movement Evoked Pain After Laparotomy for Patients With Hepatobiliary and Pancreatic Disease
Brief Title: the Effect of Doctor-nurse-patient Cooperative Analgesic Linkage Program on Movement Evoked Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2017-084
Record Dates: First submitted 2019-01-23; First posted 2019-01-31 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative; Anaplasia
Keywords: movement evoked pain; analgesia; general surgery; hepatobiliary and pancreatic disease
MeSH Terms: conditions — Pain, Postoperative; Anaplasia; Agnosia; Pancreatic Diseases | interventions — parecoxib; Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients in the experimental group were received doctor-nurse-patient cooperative analgesic linkage program.
  Interventions: Drug: Adjusted Dezocine injection; Drug: Adjusted Dynastat or Flurbiprofen Axetil jinjection; Other: postoperative rehabilitation; Drug: adjusted analgesia pump administration
- control group (Active Comparator): Patients in the control group were received routine analgesic and functional rehabilitation.
  Interventions: Drug: Routine Dezocine injection; Drug: Routine Dynastat or Flurbiprofen Axetil jinjection; Other: postoperative rehabilitation; Drug: normal analgesia pump administration

INTERVENTIONS:
Drug: Routine Dezocine injection — Dezocine 10mg were intramuscular injected at 8:00am, 4:00pm and 12:00pm.
  Other Names: Dezocine 1
  Arms: control group
Drug: Adjusted Dezocine injection — Dezocine 10mg were intramuscular injected at at 6:00am, 2:00pm and 10:00pm.
  Other Names: Dezocine 2
  Arms: Experimental Group
Drug: Routine Dynastat or Flurbiprofen Axetil jinjection — Dynastat 40mg or Flurbiprofen Axetil 50mg were administrated intravenously at 9:00am, 4:00pm and 12:00pm.
  Other Names: Dynastat or Flurbiprofen Axetil 1
  Arms: control group
Drug: Adjusted Dynastat or Flurbiprofen Axetil jinjection — Dynastat 40mg or Flurbiprofen Axetil 50mg were administrated intravenously at at 6:00am, 2:00pm and 10:00pm.
  Other Names: Dynastat or Flurbiprofen Axetil 2
  Arms: Experimental Group
Other: postoperative rehabilitation — Rehabilitation was conducted at 8:00am and 2:00pm.
  Other Names: rehabilitation
Drug: normal analgesia pump administration — Dose of analgesia pump was added if needed.
  Other Names: analgesia pump 1
  Arms: control group
Drug: adjusted analgesia pump administration — Dose of analgesia pump was added if needed. Add one dose of analgesia pump 10 minutes before rehabilitation.
  Other Names: analgesia pump 2
  Arms: Experimental Group

SUMMARY:
1. To establish doctor-nurse-patient cooperative analgesic linkage program.
2. Evaluate the effect of doctor-nurse-patient cooperative analgesic linkage program on movement evoked pain after laparotomy for patients with hepatobiliary and pancreatic disease through quasi-experimental study.

DETAILED DESCRIPTION:
Part I The establishment of doctor-nurse-patient cooperative analgesic linkage program

1. Based on literature review and clinical investigation results, initially make a doctor-nurse-patient cooperative analgesic linkage program through discussion in experts consensus meeting.
2. Using Delphi method, determine the doctor-nurse-patient cooperative analgesic linkage program after two rounds consultation.

Part II Clinical application study of doctor-nurse-patient cooperative analgesic linkage program.

Conduct non-randomized control study in corresponding period. 80 patients from two wards which managed by the same medical and nursing team were divided into experimental and control group. Patients in the control group were received routine post-operative analgesia pump and analgesics, and functional rehabilitation, while ones in the experimental group were received doctor-nurse-patient cooperative analgesic linkage program. Evaluate the effect of pain control during rehabilitation, adverse events during rehabilitation, patients' satisfaction of pain control.

ELIGIBILITY:
Inclusion Criteria:

* Consent to the study.
* Normal cognitive ability and speak Chinese
* Patients received selective laparotomy under general anesthesia.
* Length of stay is longer than three days.
* Patients who are allowed to do rehabilitation.

Exclusion Criteria:

* Patients with Severe organic disease, chronic pain, history of brain injury, history of drug or alcohol addiction.
* Psychiatric patients
* Consciousness disorder
* Patients contradict to opioid medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
movement evoked pain (Numerical rating scale) | Each rehabilitation within 3 days after surgery
  Assess movement evoked pain during rehabilitation. Numerical rating scale is a common pain rating scale. The score ranges from 0 to 10. 0 is no pain, 10 is the most severe pain.
pain at rest (Numerical rating scale) | Each rehabilitation within 3 days after surgery
  Assess pain at rest before rehabilitation.Numerical rating scale is a common pain rating scale. The score ranges from 0 to 10. 0 is no pain, 10 is the most severe pain.

SECONDARY OUTCOMES:
satisfaction questionare of pain control | three days after surgery
  Patients answer the questionare and rate the satisfaction of pain control. The questionnaire includes 7 items indicating different aspect of pain control. Patients rate their satisfaction using score. The score ranges from 1 to 5. 1 is extremely not satisfied, 5 is extremely satisfied.
the time of first bowel movement | three days after surgery
  Record the time of first bowel movement after surgery
total dose of analgesics | three days after surgery
  record and calculate the total dose of analgesics
pain at night (Numerical rating scale) | three days after surgery
  Asess the pain at rest during night.Numerical rating scale is a common pain rating scale. The score ranges from 0 to 10. 0 is no pain, 10 is the most severe pain.
adverse events during rehabilitation | three days after surgery
  adverse events during rehabilitation, such as nausea, vomiting, headache, falls

CONTACTS AND LOCATIONS:
Overall Officials: Caijuan Xu, master, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No